CLINICAL TRIAL: NCT05762315
Title: Un Protocollo di Studio Per l'Assessment Dell'Efficacia Dello Storytelling Audio Trasformativo Per Caregiver Informale (A Protocol for Assessing the Feasibility of Transformative Audio Storytelling for Informal Caregivers)
Brief Title: Transformative Audio Storytelling
Acronym: HealingStories
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Auxologico Italiano (Other)
Collaborators: European Union (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 39C101
Record Dates: First submitted 2023-02-28; First posted 2023-03-09 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Caregiver Burden
Keywords: audio storytelling; informal caregivers; digital narratives
MeSH Terms: conditions — Caregiver Burden

STUDY DESIGN:
Intervention Model Description: pre-post
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Audio Storytelling (Experimental): 15 minutes transformative audio storytelling session
  Interventions: Behavioral: Audio Storytelling

INTERVENTIONS:
Behavioral: Audio Storytelling — The audio session is designed to deliver audio narrative developed following the Transformative Storytelling Technique and provide re-structurization of internal caregiver self-stories.

SUMMARY:
Pilot testing the feasibility of the Transformative Audio Storytelling approach for informal caregivers, as an innovative method for delivering potentially empowering mental health narratives.

ELIGIBILITY:
Inclusion Criteria:

* Informal caregiver (family members or significant other person who provides primary care for the patients visiting or being hospitalized in the Rehabilitation Ward)
* Age ≥18 years
* Native speaker of the Italian language
* Having voluntarily agreed to participate in the study and having signed the informed consent in all its points.

Exclusion Criteria:

* Informal caregiver for children
* Informal caregiver who does not personally play this role (primary caregiver)
* Informal caregiver of adults with a tumor pathological condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-11-26 (Actual); Primary Completion 2022-06-10 (Actual); Study Completion 2022-09-25 (Actual)

PRIMARY OUTCOMES:
Perceived Stress Scale | pre-post (15 minutes) intervention
  The PSS is a questionnaire consisting of 10 items, on a 5-step Likert scale, ranging from 0, "Never" to 4, "Very Often". A total score of the 10 items provides a general measure of perceived stress. PPS items rate thoughts and feelings about the past month.
Sense of Coherence Scale revised (SOC-R) | pre-post (15 minutes) intervention
  The SOC-R is a tool composed of 13 items on a 5-point Likert scale ranging from 1 - "Not at all true" to 5 - "Extremely true".
Meaning in Life (MLQ) | pre-post (15 minutes) intervention
  The MLQ is a questionnaire composed of 10 items to evaluate meaning of life. The MLQ uses 7-step Likert scales from 1 "Absolutely true" to "Absolutely not true".
Cognitive Emotion Regulation Questionnaire (CERQ) | pre-post (15 minutes) intervention
  The CERQ is a questionnaire composed of 27 items, consisting of 5-step Likert scales, from 1 - "almost never" to 5 "almost always"
Facial expressions responses (Noldus FaceReader) | during 15 minutes intervention session
  this facial expression recognition software includes the evaluation of six basic expressions and then calculates the drive, valence, arousal, gaze direction, head orientation and other additional characteristics such as age and the sex
Burden Scale for Family Caregivers - Short Form (BSFC-s) | pre-post (15 minutes) intervention
  The BSFC-s is a 10-item 4-step Likert scale ranging from (0) "Strongly disagree" to (4) Strongly agree.

SECONDARY OUTCOMES:
Feedback on the perceived value of audio storytelling | after 15 minutes intervention sessions
  this facial expression recognition software includes the evaluation of six basic expressions and then calculates the drive, valence, arousal, gaze direction, head orientation and other additional characteristics such as age and the sex

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Auxologico Italiano, Milan, Lombardy, Italy